CLINICAL TRIAL: NCT00821197
Title: Long -Limb Gastric or Distal Gastric Bypass in the Treatment of Super Obese Patients - a Prospective Randomized Study
Brief Title: Long-limb or Distal Gastric Bypass for Superobesity - Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: The Hospital of Vestfold (Other)
Responsible Party: Principal Investigator, Tom Mala, Principal investigator Surgeon phd Tom Mala Rune Sandbu, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT-0910-ST
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: obesity; laparoscopy; bariatric; super obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- long-limb bypass (Active Comparator): Laparoscopic long-limb gastric bypass (150 cm alimentary limb, 50 cm biliopancreatic limb)
  Interventions: Procedure: long-limb gastric bypass
- Distal gastric bypass (Active Comparator): Laparoscopic distal gastric bypass (150 cm common channel, 50 cm biliopancreatic limb)
  Interventions: Procedure: distal gastric bypass

INTERVENTIONS:
Procedure: long-limb gastric bypass — Laparoscopic long-limb gastric bypass (150 cm alimentary limb, 50 cm biliopancreatic limb)
  Arms: long-limb bypass
Procedure: distal gastric bypass — Laparoscopic distal gastric bypass (150 cm common channel, 50 cm biliopancreatic limb)
  Arms: Distal gastric bypass

SUMMARY:
The main study objective:

To evaluate long-limb gastric bypass (150 cm alimentary limb) vs. "distal" gastric bypass (common channel 150 cm) in the treatment of superobesity (BMI 50-60 kg/m2).

The main study hypothesis:

Distal bypass accomplish an estimated 10-20 % larger weightloss than long-limb gastric bypass 1 year after surgery. Patients subject to distal bypass have more gastrointestinal side effects and more extensive nutritional deficiences compared to long-limb gastric bypass.

DETAILED DESCRIPTION:
Technical data will later be published in detail

ELIGIBILITY:
Inclusion Criteria:

* BMI 50 - 60 kg/m2 at admission for evaluation for bariatric surgery
* BMI 48 - 62 kg/m2 at study inclusion
* informed consent
* scheduled for bariatric surgery

Exclusion Criteria:

* previous bariatric surgery
* previous major abdominal surgery
* previous history or established urolithiasis
* viral hepatitis, liver cirrhosis of any kind
* factors making the patient not eligible to understand and commit to the study protocol (severe psychiatric disease or drug/narcotic abuse)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2011-02; Primary Completion 2015-05 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: weight loss | 2 years postoperatively
  physical examination

SECONDARY OUTCOMES:
Secondary outcome: Quality of life | 2 years postoperative
  questionnaire
Adverse events | 2 years postoperative
  medical history, journals
Number of patients with vitamin deficiencies | 2 years postoperative
  Blood samples
Number of patients with mineral deficiencies | 2 years postoperative
  Blood samples
Number of participants with malnutrition | 2 years postoperative
  Blood samples
Weight loss 5 year | 5 year postoperative
  physical examination
Health related Quality of life | 5 years postoperative
  questionnaire
Number of patients with malnutrition | 5 years postoperative
  Blood samples
Number of patients with mineral deficiencies | 5 years postoperative
  Blood samples
Number of patients with vitamin deficiencies | 5 years postoperative
  Blood samples
Adverse events | 5 years
  Medical history, journals
Weight loss 10 years | 10 years postoperative
  Weight measure
Adverse events | 10 years postoperative
  Medical history, journals
Number of patients with malnutrition | 10 years postoperative
  Blood samples
Number of patients with mineral deficiencies | 10 years postoperative
  Blood samples
Number of patients with vitamin deficiencies | 10 years postoperative
  Blood samples
Health related Quality of life | 10 years postoperative
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tom Mala MD, PhD Rune Sandbu, MD, PhD, Study Chair — Aker University Hospital / The Hospital of Vestfold
Locations (1):
- Aker university Hospital, Surgical Dep., The Hospital of Vestfold, Surgical Dep., Oslo, Norway

REFERENCES:
- [Derived] Salte OB, Hagen RE, Svanevik M, Fagerland MW, Risstad H, Hjelmesaeth J, Kristinsson JA, Sandbu R, Mala T. Effect of standard versus long alimentary limb distal Roux-en-Y gastric bypass on weight loss and nutritional outcomes at 10 years in patients with BMI 50-60 kg/m2-a secondary analysis of a randomized clinical trial. Br J Surg. 2025 Dec 24;113(1):znaf285. doi: 10.1093/bjs/znaf285. PMID 41553109
- [Derived] Salte OBK, Svanevik M, Risstad H, Hofso D, Blom-Hogestol IK, Johnson LK, Fagerland MW, Kristinsson J, Hjelmesaeth J, Mala T, Sandbu R. Standard versus distal Roux-en-Y gastric bypass in patients with BMI 50-60 kg/m2: 5-year outcomes of a double-blind, randomized clinical trial. BJS Open. 2021 Nov 9;5(6):zrab105. doi: 10.1093/bjsopen/zrab105. PMID 34791048
- [Derived] Svanevik M, Risstad H, Hofso D, Blom-Hogestol IK, Kristinsson JA, Sandbu R, Smastuen MC, Thorsby PM, Mala T, Hjelmesaeth J. Bone Turnover Markers After Standard and Distal Roux-en-Y Gastric Bypass: Results from a Randomized Controlled Trial. Obes Surg. 2019 Sep;29(9):2886-2895. doi: 10.1007/s11695-019-03909-1. PMID 31065919
- [Derived] Svanevik M, Risstad H, Karlsen TI, Kristinsson JA, Smastuen MC, Kolotkin RL, Sovik TT, Sandbu R, Mala T, Hjelmesaeth J. Patient-Reported Outcome Measures 2 Years After Standard and Distal Gastric Bypass-a Double-Blind Randomized Controlled Trial. Obes Surg. 2018 Mar;28(3):606-614. doi: 10.1007/s11695-017-2891-3. PMID 28865057
- [Derived] Risstad H, Svanevik M, Kristinsson JA, Hjelmesaeth J, Aasheim ET, Hofso D, Sovik TT, Karlsen TI, Fagerland MW, Sandbu R, Mala T. Standard vs Distal Roux-en-Y Gastric Bypass in Patients With Body Mass Index 50 to 60: A Double-blind, Randomized Clinical Trial. JAMA Surg. 2016 Dec 1;151(12):1146-1155. doi: 10.1001/jamasurg.2016.2798. PMID 27626242
- [Derived] Svanevik M, Risstad H, Hofso D, Schou CF, Solheim B, Sovik TT, Kristinsson J, Hjelmesaeth J, Mala T, Sandbu R. Perioperative Outcomes of Proximal and Distal Gastric Bypass in Patients with BMI Ranged 50-60 kg/m(2)--A Double-Blind, Randomized Controlled Trial. Obes Surg. 2015 Oct;25(10):1788-95. doi: 10.1007/s11695-015-1621-y. PMID 25761943
- See also: hospital site — http://www.aus.no/
- See also: hospital site — http://www.siv.no